CLINICAL TRIAL: NCT07169370
Title: SPIRIT Club CBI Pathway: A Novel Streaming Platform for Physical Activity and Wellness Promotion for Chronic Brain Injury Survivors
Brief Title: SPIRIT Club Chronic Brain Injury Exercise Platform
Acronym: SPIRITClubCBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine Quatman-Yates, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024H0167; R44HD112248 (NIH)
Record Dates: First submitted 2025-08-28; First posted 2025-09-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Brain Injury
Keywords: fitness platform; chronic brain injury
MeSH Terms: conditions — Brain Injury, Chronic

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-assignment, single-masked interventional study with two arms:
  Intervention Arm: Participants receive access to the SPIRIT Club CBI Pathway streaming platform and a Fitbit for continuous activity monitoring.
  Control Arm: Participants receive a Fitbit alone, plus weekly check-ins, but no platform access.
  Participants are randomized 1:1 and followed for 8 weeks. Outcome assessors remain masked to arm assignment. Primary feasibility and activity outcomes (e.g., tracked activity, exercise self-efficacy) are measured at baseline and week 8.
Who Masked: Outcomes Assessor
Masking Description: The investigators operationally define 'Outcomes Assessor' for this trial as the biostatistician, who will be unaware of participant group assignments during the final data analysis.
  The data for key outcomes, such as feasibility and acceptability, are generated directly by the participants themselves through their survey responses and interaction with the platform.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIRIT Club CBI Pathway (Experimental): Participants receive free, two-month access to the SPIRIT Club CBI Pathway on-demand streaming platform, featuring targeted educational modules and adaptive exercise programming designed specifically for CBI survivors and their caregivers, plus a Fitbit Inspire 3 to wear continuously for the purposes of activity monitoring over the intervention period.
  Interventions: Behavioral: SPIRIT Club CBI Pathway
- Activity Monitoring Only (No Intervention): There is no intervention in this Arm. In order to track activity, participants will undergo the same activity monitoring procedures as the experimental group.

INTERVENTIONS:
Behavioral: SPIRIT Club CBI Pathway — A tailored, on-demand exercise and education program delivered via the SPIRIT Club virtual streaming platform. Content includes progressive adaptive workouts, safety videos, screening checkpoints, and prompts for a support person. Participants choose classes designed specifically for adults ≥9 months post-brain injury and after being placed in the appropriate archetype, complete activity surveys, and earn incentives for adherence. They are instructed on current physical activity guidelines (≥150 min moderate or ≥75 min vigorous activity per week) and to follow the CBI Pathway at their comfort level. Content was co-developed with clinical experts and survivors to ensure both usability and safety.
  Other Names: CBI Pathway; SPIRIT Club streaming fitness platform
  Arms: SPIRIT Club CBI Pathway

SUMMARY:
Many physical fitness centers and online exercise programs are not designed to support people with intellectual and developmental disabilities. To address this, the investigators are collaborating with SPIRIT Club, a company specializing in fitness for people with disabilities, to improve their platform. The goal is to create a new section of the platform specifically for people with chronic brain injury (CBI). The investigators will test and refine this new section to see how well it works for people with CBI in real-life situations. The research will focus on conducting a study with 60 people who have CBI to see if the new section helps them be more active and confident in their ability to exercise. Half will use the new section, and the other half will just be monitored for their activity. The investigators includes experts in fitness and rehabilitation for people with disabilities from industry, clinical settings, and research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older with chronic brain injury (CBI)
* At least 9 months post-injury
* Is able to able to be able to demonstrate the ability to meet at least one of the following functional mobility scenarios: 1) able to walk with or without an assistive device or with no more than contact guard assist from a caregiver for steadiness checks and proprioceptive support, 2) able to stand up from a chair with no assistance or no more than contact guard assist from a caregiver for steadiness and proprioceptive support, and/or 3) able to maintain steady seated balance in a chair or wheelchair and able to lift at least one limb with minimal assist (<25%) from a caregiver against gravity
* Currently exercising less than 60 minutes per week
* Able to follow simple commands
* Participant is his/her own legal authorized representative (LAR) or LAR is able to verify they can follow simple commands and participate in study and support consenting and participation processes
* Provides confirmation of medical clearance from physician to participate in moderate levels of activity without supervision from a licensed healthcare provider

Exclusion Criteria:

* Unsafe independent functional mobility observed during the functional mobility screen and no available caregiver/carepartner to facilitate participation in the study and provide assistance while using the SPIRIT Club platform
* Being advised by any healthcare provider to avoid or restrict participation in moderate to high-intensity physical activity
* Uncontrolled blood pressure, unstable angina, severe joint disease, uncontrolled or untreated dizziness or vertigo, or other medical issue precluding exercises leading to lack of clearance from a physician
* - e.g.,
* Unable to follow simple commands or persistent post-traumatic amnesia
* Presence of expressive aphasia
* Lack of fluency in English
* Unable to follow simple commands or persistent post-traumatic amnesia
* Regular participation (2 or more days per week) in a structured fitness program or platform (e.g., group exercise classes or personal training)
* Regular participation (average of 1 or more days per week) in physical therapy services specifically for brain injury rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From enrollment through completion of the intervention (Week 8).
  Feasibility will be assessed over the intervention period using recruitment rate (number of enrolled participants relative to those approached) as an objective indicator.
Attendance of SPIRIT Club CBI Pathway Sessions | From enrollment through completion of the intervention (Week 8).
  Feasibility will be assessed over the intervention period using attendance (number of sessions completed) as an objective indicator.
Attrition Rate | From enrollment through completion of the intervention (Week 8).
  Feasibility will be assessed over the intervention period using attrition rate (proportion withdrawing before end of the intervention period as an objective indicator.
Unplanned Study-team contacts during enrollment | From enrollment through completion of the intervention (Week 8).
  Feasibility will be assessed over the intervention period using unplanned study-team contacts (number of emails and/or calls outside scheduled check-ins; total and per participant) as an objective indicator.
Accessibility Issues | From enrollment through completion of the intervention (Week 8).
  Feasibility will be assessed over the intervention period using accessibility issues (number of instances where participants could not successfully acquire or use the streaming platform or data-collection tools; participant and/or staff team reported) as an objective indicator.
Safety of the SPIRIT Club CBI Pathway Platform | From enrollment through completion of the intervention (Week 8).
  Safety will be assessed through the documentation of exercise-related adverse events (number per participant and total over the intervention period).
Acceptability Survey | At program end (Week 8).
  Acceptability will be evaluated immediately after the 8-week program or at the time of withdrawal using an electronically administered survey. The investigators will assess acceptability based on answers to a 5-point satisfaction scale (1 = very dissatisfied to 5 = very satisfied) for (1) overall program content and (2) usability and a series of binary yes/no responses to the following questions: "Was the program worth the participant's time?" and "Would the participant recommend it to others with CBI?"; and open-ended comments capturing likes, dislikes, and improvement suggestions.
Exercise Self-Efficacy Scale Score | Baseline and Week 8
  Electronic survey administered to participant. Change in total score on the validated 6-item exercise self-efficacy scale, from baseline to Week 8, which assesses participants' confidence to engage in physical activity despite common barriers.

SECONDARY OUTCOMES:
Step Count | From enrollment through completion of the intervention (Week 8).
  Activity is monitored using a Fitbit Inspire 3 wearable device, which captures daily step count.
Active Minutes | From enrollment through completion of the intervention (Week 8).
  This outcome provides a comprehensive assessment of participants' physical activity patterns by a Fitbit Inspire 3 wearable device, which captures active minutes in intensity zones.
Platform Utilization - Total Classes Initiated | Weekly summaries during Weeks 1-8.
  Utilization metrics will be drawn from the SPIRIT Club streaming platform's automatic logs on a weekly basis (Weeks 1-8), including total number of classes initiated These data quantify how frequently and intensively participants engage with the CBI Pathway.
Platform Utilization - Minutes of Video Streamed | Weekly summaries during Weeks 1-8.
  Utilization metrics will be drawn from the SPIRIT Club streaming platform's automatic logs on a weekly basis (Weeks 1-8), including cumulative minutes of video streamed (group total and per participant).
Daily Activity Log - Tracked Activity Counts | From enrollment through completion of the intervention (Week 8)
  The total number of activities completed each day, as measured by a participant-completed daily activity log.
Daily Activity Log - Tracked Activity Minutes | From enrollment through completion of the intervention (Week 8).
  The total duration of activity in minutes each day, as measured by a participant-completed daily activity log.

OTHER OUTCOMES:
Health-Promoting Lifestyle Profile II (HPLP II) Physical Activity Domain | Baseline and Week 8
  Electronic survey administered to participant. Change in total score on the validated 8-item questionnaire, from baseline to Week 8, that assesses the extent to which an individual engages in a health-promoting lifestyle, specifically with physical activity. For each item, participants rate how often they engage in the described behavior on a 4-point scale (1=Never, 2=Sometimes, 3=Often, 4=Routinely). Total scores are calculated by summing the responses, with higher scores indicating a more health-promoting lifestyle.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
To protect the privacy and confidentiality of our study participants, individual participant data (IPD) will not be shared.

REFERENCES:
- See also: Official homepage for SPIRIT Club, a virtual on-demand fitness streaming platform offering adaptive, progressive exercise classes and educational modules for people with disabilities, including those with chronic brain injury. — https://www.spirit-club.com/